CLINICAL TRIAL: NCT03758404
Title: An Open Label, Multi-centre, Phase I/II Dose Escalation Trial of a Recombinant Adeno-associated Virus Vector (AAV2/8-hG1.7p.coCNGA3) for Gene Therapy of Children and Adults With Achromatopsia Owing to Defects in CNGA3
Brief Title: Gene Therapy for Achromatopsia (CNGA3)
Acronym: CNGA3
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MeiraGTx UK II Ltd (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MGT012
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Results first posted 2022-02-11 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Achromatopsia
MeSH Terms: conditions — Color Vision Defects

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low dose adeno-associated virus (AAV) CNGA3 (Experimental): Subretinal administration of a single low dose AAV CNGA3
  Interventions: Biological: adeno-associated virus vector AAV- CNGA3
- Intermediate dose adeno-associated virus (AAV) CNGA3 (Experimental): Subretinal administration of a single intermediate dose AAV CNGA3
  Interventions: Biological: adeno-associated virus vector AAV- CNGA3
- High dose adeno-associated virus (AAV) CNGA3 (Experimental): Subretinal administration of a single high dose AAV CNGA3
  Interventions: Biological: adeno-associated virus vector AAV- CNGA3

INTERVENTIONS:
Biological: adeno-associated virus vector AAV- CNGA3 — Adeno-associated virus (AAV) gene therapy for defects in CNGA3 gene

SUMMARY:
A clinical trial of adeno-associated virus vector (AAV) CNGA3 retinal gene therapy for patients with achromatopsia

DETAILED DESCRIPTION:
CNGA3 retinal gene therapy for patients with achromatopsia

ELIGIBILITY:
Inclusion Criteria:

* Are aged years or over
* Have achromatopsia confirmed by a retinal specialist investigator

Exclusion Criteria:

* Are females who are pregnant or breastfeeding
* Have participated in another research study involving an investigational medicinal therapy for ocular disease within the last 6 months
* Have any other condition that the investigator considers makes them inappropriate for entry into the trial

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Bainbridge, Principal Investigator — Chief Investigator
Locations (2):
- Kellogg Eye Center, Ann Arbor, Michigan, United States
- Moorfields Eye Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from two medical centers between 12 August 2019 (date first participant signed informed) and 19 November 2020 (date last participant signed informed consent). A total of 11 participants were enrolled in the study.
Groups:
- Low Dose AAV - CNGA3: Subretinal administration of a single low dose adeno-associated virus AAV-CNGA3
  AAV-CNGA3: AAV gene therapy for defects in CNGA3 gene
- Intermediate Dose AAV - CNGA3: Subretinal administration of a single intermediate dose adeno-associated virus AAV-CNGA3
  AAV- CNGA3: AAV gene therapy for defects in CNGA3 gene
- High Dose AAV - CNGA3: Subretinal administration of a single high dose adeno-associated virus AAV-CNGA3
  AAV- CNGA3: AAV gene therapy for defects in CNGA3 gene
Period: Overall Study
Arm/Group | Low Dose AAV - CNGA3 | Intermediate Dose AAV - CNGA3 | High Dose AAV - CNGA3
Started | 3 | 3 | 5
Completed | 3 | 3 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Low Dose AAV - CNGA3: Subretinal administration of a single low dose AAV - CNGA3
  AAV- CNGA3: AAV gene therapy for defects in CNGA3 gene
- Intermediate Dose AAV - CNGA3: Subretinal administration of a single intermediate dose AAV - CNGA3
  AAV- CNGA3: AAV gene therapy for defects in CNGA3 gene
- High Dose AAV - CNGA3: Subretinal administration of a single high dose AAV - CNGA3
  AAV- CNGA3: AAV gene therapy for defects in CNGA3 gene
- Total: Total of all reporting groups
Arm/Group | Low Dose AAV - CNGA3 | Intermediate Dose AAV - CNGA3 | High Dose AAV - CNGA3 | Total
Number analyzed (Participants) | 3 | 3 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 3 | 3 | 9
  Between 18 and 65 years | 0 | 0 | 2 | 2
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 2
  Male | 2 | 3 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 3 | 3 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 1 | 2 | 3 | 6
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 0 | 0 | 2 | 2
  United Kingdom | 3 | 3 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Meeting the Primary Outcome Defined as Any of the Below Events Occurring During the 6 Weeks Following Administration, at Least Possibly Related to the Advanced Therapy Investigational Medicinal Products (ATIMP), Not Surgery Alone.
Description: The primary outcome is defined as any of the below occurring during the 6 weeks following administration, at least possibly related to the Advanced Therapy Investigational Medicinal Products (ATIMP), not surgery alone:
  * Reduction in visual acuity by 15 Early Treatment Diabetic Retinopathy Study (ETDRS) letters or more that fails to resolve to within 15 letters of baseline in a 4-week period once prophylactic treatment commences
  * Severe unresponsive inflammation
  * Infective endophthalmitis
  * Ocular malignancy
  * Grade III or above non-ocular Suspected Unexpected Serious Adverse Reaction (SUSAR)
Time Frame: 6 Weeks
Population: The safety analysis set included all enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose AAV - CNGA3 | Intermediate Dose AAV - CNGA3 | High Dose AAV - CNGA3
Number analyzed (Participants) | 3 | 3 | 5
Participants | 0 | 0 | 0

2. Secondary Outcome: Improvements in Visual Function as Assessed by Visual Acuity
Description: Change from baseline to Week 24 in best corrected visual acuity (BCVA) using Early Treatment Diabetic Retinopathy Study (ETDRS) chart letter score. The direction of improvement from baseline is an increase in the number of ETDRS letters read over time.
Time Frame: 6 Months
Population: All of the 11 participants performed the visual acuity assessment at baseline and Week 24.
Measure: Mean (Full Range); unit: number of ETDRS letters
Groups:
- Overall: Subretinal administration of a single low, intermediate, or high dose AAV CNGA3
  adeno-associated virus vector AAV- CNGA3: Adeno-associated virus (AAV) gene therapy for defects in CNGA3 gene
Arm/Group | Low Dose Adeno-associated Virus (AAV) CNGA3 | Intermediate Dose Adeno-associated Virus (AAV) CNGA3 | High Dose Adeno-associated Virus (AAV) CNGA3 | Overall
Number analyzed (Participants) | 3 | 3 | 5 | 11
number of ETDRS letters | 0.22 [-0.7 to 1.3] | 2.44 [0.0 to 4.7] | 2.40 [-1.0 to 5.0] | 1.82 [-1.0 to 5.0]

3. Secondary Outcome: Improvements in Retinal Function as Assessed by Static Perimetry
Description: Change from baseline to Week 24 in mean retinal sensitivity in the treated eye. The direction of improvement is an increase in sensitivity.
Time Frame: 6 Months
Population: Six of the 11 participants had mean retinal sensitivity data available at both baseline and Week 24 in the treated eye.
Measure: Mean (Full Range); unit: decibel
Arm/Group | Low Dose Adeno-associated Virus (AAV) CNGA3 | Intermediate Dose Adeno-associated Virus (AAV) CNGA3 | High Dose Adeno-associated Virus (AAV) CNGA3 | Overall
Number analyzed (Participants) | 1 | 1 | 4 | 6
decibel | 1.17 | -1.83 | 0.15 [-0.3 to 0.9] | -0.01 [-1.8 to 1.2]

4. Secondary Outcome: Quality of Life Measured by QoL Questionnaires in Children and Adolescents
Description: Change from baseline to Week 24 in EuroQol Visual Analogue Scale (EQ-VAS) in children and adolescents. EQ-VAS uses a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state. A positive change from baseline reflects improvement and a negative reflects worsening.
Time Frame: 6 Months
Population: EQ-VAS data were available for 6 of the 9 children/adolescents enrolled in the study.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Low Dose Adeno-associated Virus (AAV) CNGA3 | Intermediate Dose Adeno-associated Virus (AAV) CNGA3 | High Dose Adeno-associated Virus (AAV) CNGA3 | Overall
Number analyzed (Participants) | 1 | 3 | 2 | 6
units on a scale | -15 | 18.3 [-1 to 50] | 8.0 [0 to 16] | 9.3 [-15 to 50]

5. Secondary Outcome: Quality of Life Measured by QoL Questionnaires in Adults
Description: Change from baseline to Week 24 in EuroQol Visual Analogue Scale (EQ-VAS) in adults. EQ-VAS uses a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state. A positive change from baseline reflects improvement and a negative reflects worsening.
Time Frame: 6 Months
Population: EQ-VAS data were available for both adults enrolled in the study.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Low Dose Adeno-associated Virus (AAV) CNGA3 | Intermediate Dose Adeno-associated Virus (AAV) CNGA3 | High Dose Adeno-associated Virus (AAV) CNGA3 | Overall
Number analyzed (Participants) | 0 | 0 | 2 | 2
units on a scale |  |  | 1.5 [-7 to 10] | 1.5 [-7 to 10]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Low Dose AAV - CNGA3 | Intermediate Dose AAV - CNGA3 | High Dose AAV - CNGA3
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose AAV - CNGA3 (N=3) | Intermediate Dose AAV - CNGA3 (N=3) | High Dose AAV - CNGA3 (N=5)
Conjunctival haemorrhage (Eye disorders) | 3 | 3 | 5
Visual acuity reduced (Eye disorders) | 3 | 3 | 2
Conjunctival hyperaemia (Eye disorders) | 1 | 3 | 2
Lenticular opacities (Eye disorders) | 1 | 3 | 2
Ocular discomfort (Eye disorders) | 1 | 1 | 4
Eye inflammation (Eye disorders) | 0 | 0 | 2
Eye pain (Eye disorders) | 1 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 2
Subconjunctival cyst (Eye disorders) | 0 | 1 | 1
Chorioretinal folds (Eye disorders) | 0 | 0 | 1
Foreign body sensation in eyes (Eye disorders) | 0 | 1 | 0
Iridocyclitis (Eye disorders) | 0 | 0 | 1
Photophobia (Eye disorders) | 1 | 0 | 0
Punctate keratitis (Eye disorders) | 0 | 1 | 0
Retinal disorder (Eye disorders) | 0 | 0 | 1
Uveitis (Eye disorders) | 0 | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 1 | 0
Intraocular pressure increased (Investigations) | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 1
Intraocular pressure decreased (Investigations) | 1 | 0 | 0
Slit-lamp tests abnormal (Investigations) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperlipidaemia (Endocrine disorders) | 0 | 0 | 1
Type 2 diabetes mellitus (Endocrine disorders) | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 0
Tenon's cyst (Injury, poisoning and procedural complications) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-04-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT03758404/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/04/NCT03758404/SAP_001.pdf